CLINICAL TRIAL: NCT04669990
Title: Remdesivir and Convalescent Plasma Therapy for Treatment of COVID-19 Infection in Nepal : A Registry Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nepal Health Research Council (Other Government)
Responsible Party: Principal Investigator, Dr. Pradip Gyanwali,MD, Member-Secretary, Nepal Health Research Council
Other Study IDs: 749-2020
Record Dates: First submitted 2020-12-14; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — remdesivir

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Drug: Remdesivir — The objective of this Registry study is to continue to collect safety and outcome data for COVID-19 patients who are treated with Remdesivir and convalescent plasma therapy (CPT).
  Other Names: Convalescent Plasma

SUMMARY:
The pandemic COVID-19 does not have an established treatment. Clinical trials of antiviral drugs against SARS CoV-2 are currently in progress. Clinical study done by NIH which included 1059 patients indicated that those who received Remdesivir had a median recovery time of 11 days as compared with 15 days in those who received placebo. Remdesivir has recently received full approval for COVID-19 by US FDA, and emergency use authorization (EUA) by multiple countries including European Commission and Indian Health Service. Remdesivir appears to demonstrate the most benefit in those with severe COVID-19 on supplemental oxygen. The NIH Panel recommends using Remdesivir for 5 days or until hospital discharge, whichever comes first. The interim analysis of WHO's SOLIDARITY trial, however, failed to show mortality benefit with Remdesivir. Review of literature suggests the transfusion of convalescent plasma has been used successfully in observational and retrospective studies. A recent metanalysis showed that convalescent plasma reduced mortality by 57% compared to matched-patients receiving standard treatments. The objective of NHRC sponsored initial clinical study protocol (Convalescent Plasma study) was to provide a coordinated approach for collection and preparation, distribution and guidance for safe and effective administration of convalescent plasma with antibodies against SAR CoV-2 for treatment of patients with COVID-19 infection who are most likely to benefit from this investigational treatment. On August 9th, 2020, the Government of Nepal gave permission to use Remdesivir in COVID-19 patients of Nepal only as a study drug when the original protocol was amended to add a second study arm to use Remdesivir for treatment of patients with moderate to severe COVID-19. The enrollment goal of these two protocols have been reached and collection of study data will be completed by the end of October 2020. On October 18th, the GoN MoHP also announced and directed to provide access for Remdesivir directly through the pharmacies. Therefore, this registry study has been designed to replace the compassionate use study of Remdesivir and Convalescent plasma.

DETAILED DESCRIPTION:
The pandemic COVID-19 does not have an established treatment. Although small studies have demonstrated some successes of few antiviral and immunomodulatory agents, either their data so far are not very encouraging (e.g. Hydroxychloroquine and Antiretroviral Protease Inhibitors) or clinical trials of newly introduced drugs are currently in progress and not available in Nepal. Review of literature suggests the transfusion of convalescent plasma has been used successfully in small observational and retrospective studies. A recent metanalysis showed that convalescent plasma reduced mortality by 57% compared to matched-patients receiving standard treatments. While multiple antiviral drugs are undergoing clinical trials and there is no established antiviral agents against COVID-19, the infectious diseases guidelines suggest use of Remdesivir among hospitalized patients with severe COVID-19 patients (Conditional recommendation, moderate certainty of evidence). Clinical study done by NIH which included 1059 patients indicated that those who received Remdesivir had a median recovery time of 11 days as compared with 15 days in those who received placebo. Remdesivir has received emergency use authorization for COVID-19 by US FDA, European Commission, and Indian Health Service. Remdesivir appears to demonstrate the most benefit in those with severe COVID-19 on supplemental oxygen. The NIH Panel recommends using Remdesivir for 5 days or until hospital discharge, whichever comes first. The interim analysis of WHO's SOLIDARITY trial, however, failed to show mortality benefit with Remdesivir.The objective of initial clinical protocol (Convalescent Plasma study) was to provide a coordinated approach for collection and preparation, distribution and guidance for safe and effective administration of convalescent plasma with antibodies against SAR CoV-2 for treatment of patients with COVID-19 infection who are most likely to benefit from this investigational treatment. On August 9th, 2020, the Government of Nepal gave permission to use Remdesivir in COVID-19 patients of Nepal only as a study drug when the original protocol was been amended to add a second study arm for use of Remdesivir for treatment of patients with moderate to severe COVID-19. The enrollment goal of these two protocols have been reached and collection of study data will be completed by the end of October 2020. On October 18th, the GoN MoHP also announced and directed to provide access for Remdesivir directly through the pharmacies. Therefore, this registry study has been designed to replace the compassionate use study of Remdesivir and Convalescent plasma.

ELIGIBILITY:
Inclusion Criteria:

* All patients who receive treatment with CPT or Remdesivir will be eligible for the study. Treatment decision will be based on decision of the treating physicians. However, following guidelines for treatment are provided based on current standard of care: For Remdesivir: Patients with severe COVID-19 infection who require to be on oxygen supplementation.

For convalescent plasma therapy: Patients who meet one of the following criteria are likely to benefit from convalescent plasma therapy:

1. Patients on life-threatening COVID-19 infection when combined with Remdesivir.
2. Patients who progress to life-threatening infection despite being on remdesivir for 48 hours or longer. The following definitions are used to define severe and life threatening COVID-19 infection.

Severe COVID-19 infection is defined by one or more of the following criteria:

1. Shortness of breath (dyspnea)
2. Respiratory frequency ≥ 30/min
3. Blood oxygen saturation ≤ 93%
4. Partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300
5. Lung infiltrates increased more than 50% within 24 to 48 hours

Life-threatening COVID-19 infection is defined as one or more of the following:

1. Respiratory failure
2. Septic shock
3. Multiple organ dysfunction or failure

Exclusion Criteria:

1. If the diagnosis is not confirmed with PCR or similar alternative tests for COVID-19 infection
2. Any patient with contraindications for receiving plasma transfusion should not receive plasma
3. Any patient with contraindications for receiving Remdesivir should not receive Remdesivir

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from all COVID-19 treating hospitals of Nepal which are participating in this clinical study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-11-19 (Estimated)

PRIMARY OUTCOMES:
Demographics of recipients | 9 Months
  - type of patients receiving plasma therapy : Age in Years, Sex: M/F
Co-morbidity of recipient | 9 Months
  - recipient comorbidities: Smoking, Diabetes, Heart disease, Chronic lung disease, chronic liver disease, cancer, organ transplant, HIV infection, TB. HIV, HBV, HCV, Syphillis
Adverse events of convalescent COVID-19 plasma and Remdesivir Therapy | 9 Months
  * any expected and unexpected adverse events during or after treatment (upto 7 days)
  * any other complications related or unrelated to plasma transfusion and Remdesivir during hospital stay
Hospital and ICU length of stay | 9 Months
  - number of days of hospital stay and ICU stay
Disposition of patients including survival | 9 Months
  - condition at discharge: complete recovery, partial recovery with complications, death

CONTACTS AND LOCATIONS:
Locations (4):
- Nepal (4):
  - Narayani Hospital, Birgunj
  - Seti Provincial Hospital, Dhangadi
  - BP Koirala Institute of Health Sciences (BPKIHS), Dharān
  - Bheri Provincial Hospital, Nepalgunj